CLINICAL TRIAL: NCT06281977
Title: Study Evaluating Dexmedetomidine in the Acute Treatment of Electrical Storm
Acronym: SEDATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ES613
Record Dates: First submitted 2024-02-09; First posted 2024-02-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Ventricular Tachycardia; Ventricular Arrhythmias; Ventricular Fibrillation; Recurrent Ventricular Tachycardia
Keywords: Electrical Storm; Dexmedetomidine; Ventricular Electrical Storm; Precedex; Recurrent Ventricular Arrhythmias; Recurrent Ventricular Tachycardia; Sedation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Participants randomized to receive dexmedetomidine will be started at a dose of 0.3 mcg/kg/hr and titrated to a target dose of 1.0 mcg/kg/hr. Once the participant reaches their maximum tolerated dose (as decided by the blinded treating physician), they will continue treatment for 48 ± 6 hours. This will be followed by a weaning phase that will similarly be at the discretion of the treating physician.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Participants randomized to receive placebo will be started on normal saline. In similar fashion to the active comparator, participants will be titrated to their maximal tolerated dose, continue treatment for 48 ± 6 hours, and be weaned at the discretion of the blinded treating physician.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dose range: 0.3 mcg/kg/hr to 1 mcg/kg/hr.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Normal saline — Programed as dexmedetomidine on infusion pump.
  Arms: Placebo

SUMMARY:
The objective of this study is to determine if there is a meaningful benefit to using the sedative medication dexmedetomidine in the acute treatment of patients with recurrent ventricular arrhythmias, known as electrical storm. This will be a multi-centre, double-blinded, placebo-controlled, randomized trial. Patients with electrical storm will be randomized to receive 48 to 72 hours of dexmedetomidine or placebo as part of their initial treatment in an intensive care unit.

DETAILED DESCRIPTION:
Electrical storm (ES), defined as three or more sustained or treated ventricular arrhythmias in a 24-hour period, is a life-threatening condition that is associated with significant short- and long-term mortality. Autonomic dysfunction from increased sympathetic tone and the catecholamine surge from defibrillator shocks can precipitate recurrent ventricular arrhythmias and exacerbate ES. Although the mainstay of treatment are anti-arrhythmic drugs, sedative agents and procedures are commonly used to decrease sympathetic tone. These therapies have been studied in refractory ES but the benefit of early sedation remains unclear.

Alpha-2 agonism with dexmedetomidine can provide conscious sedation without the need for mechanical ventilation. Dexmedetomidine has been found to reduce ventricular arrhythmia events in non-ES patients in the intensive care unit and in the peri-operative period. Its antiarrhythmic properties are thought to be due to catecholamine suppression, prolonging electrical refractory periods, and increasing vagal tone. Its rapid onset and favorable safety profile render alpha-2 agonism with dexmedetomidine a potentially valuable therapy for patients with ES.

This study is a multi-centre, double-blinded, placebo-controlled, randomized trial that will evaluate the effectiveness of dexmedetomidine in the acute treatment of ES. Consecutive patients admitted to an intensive care unit will be randomized to receive dexmedetomidine or placebo at the time of presentation. The study drug will be titrated to a maintenance dose and continued for 48 hours before being weaned.

ELIGIBILITY:
Inclusion Criteria:

- All patients admitted to an intensive care unit with electrical storm over the age of 18 years will be approached for enrollment.

Exclusion Criteria:

* Refractory shock lasting for more than 30 minutes unrelated to ventricular arrhythmias (VAs), defined as requiring two or more vasopressors
* SCAI class D or E cardiogenic shock
* Cardiac arrest(s) with a no-flow and low-flow total time of greater than 10 minutes prior to recruitment.
* ST-segment elevation myocardial infarction (STEMI)-induced VA with signs of active ischemia.
* Bradycardia with heart rate less than 40 beats per minute, bradycardia-induced ventricular tachyarrhythmia, second degree Mobitz type 2 or greater atrioventricular block in the absence of a pacemaker.
* Pregnancy
* Known dexmedetomidine allergy or intolerance
* Inability to obtain consent from patient or substitute decision maker.
* Patients who have received dexmedetomidine or clonidine during the 24 hours prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 192 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-05-08 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is a composite of the following: 1. All-cause in-hospital death AND/OR 2. Any in-hospital ventricular arrhythmia requiring treatment after study drug initiation. | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo

SECONDARY OUTCOMES:
All-cause in-hospital death | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Ventricular arrhythmia requiring treatment after study drug initiation | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Resuscitated cardiac arrest after study drug initiation | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Renal failure requiring new initiation of renal replacement therapy after study drug initiation | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Intubation following study drug initiation | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Length of stay in the intensive care unit | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Length of stay in hospital | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Need for mechanical circulatory support device after study drug initiation | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo
Ventricular Arrhythmia requiring treatment only during active study drug treatment | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime the participant is receiving dexmedetomidine or normal saline placebo
Pacing or treatment with isoproterenol for treatment of bradyarrhythmia after study drug initiation. | Duration of index hospitalization - an average of 2 weeks
  Defined as anytime after the participant starts receiving dexmedetomidine or normal saline placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study data, protocol, SAP, ICF, and CSR will be made available at study completion/publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study completion
Access Criteria: The above will be made publicly available

REFERENCES:
- [Derived] Motazedian P, Santo PD, Prosperi-Porta G, Nelson D, Morgan B, Ratelle C, Feagan H, Koopman Z, Jung R, Mathieu ME, Knoll W, Parlow S, Abdel-Razek O, Mathew R, Wells GA, Chiu MH, Ballantyne B, Hibbert B, Ramirez FD. Study Evaluating Dexmedetomidine in the Acute Treatment of Electrical storm (SEDATE): rationale and design. Am Heart J. 2026 Jan 25:107358. doi: 10.1016/j.ahj.2026.107358. Online ahead of print. PMID 41592634